CLINICAL TRIAL: NCT01162746
Title: Comparison of Intravitreal Dexamethasone With Intravitreal Ranibizumab Versus Intravitreal Ranibizumab Monotherapy in Recurrent or Persistent Choroidal Neovascularization Secondary to Age-related Macular Degeneration A Prospective, Randomized, Clinical Study
Brief Title: Comparison of Ranibizumab Monotherapy and Ranibizumab Combination Therapies in Recurrent or Persistent Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Ass.-Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10032011
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Age-Related Macular Degeneration; Neovascularization, Choroidal
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Intravitreal dexamethasone and intravitreal ranibizumab (Experimental): Patients will receive intravitreal dexamethasone using a special drug delivery system and same day intravitreal ranibizumab.
  Study medications are initially given at the baseline visit. At each subsequent monthly follow-up visit, ranibizumab is administered if further visual deterioration or persistence of sub-/intraretinal fluid is detected in the examination. At month 3, 6, 9 and 12 further treatments with intravitreal dexamethasone in combination with intravitreal ranibizumab are given if leakage is detected in fluorescein or indocyanine green (FLA or ICG) angiography, in case of further vision decrease or persistence of sub-/intraretinal fluid in OCT.
  Interventions: Drug: Intravitreal dexamethasone and intravitreal ranibizumab
- Intravitreal ranibizumab (Active Comparator): Patients will receive intravitreal ranibizumab monotherapy (cohort 3). Study medications are initially given at the baseline visit. At each subsequent monthly follow-up visit, ranibizumab is administered if further visual deterioration or persistence of sub-/intraretinal fluid is detected in the examination
  Interventions: Drug: Intravitreal ranibizumab

INTERVENTIONS:
Drug: Intravitreal dexamethasone and intravitreal ranibizumab — Patients will receive intravitreal dexamethasone using a special drug delivery system and same day intravitreal ranibizumab.
  Study medications are initially given at the baseline visit. At each subsequent monthly follow-up visit, ranibizumab is administered if further visual decrease or persistence of sub-/intraretinal fluid is detected in the examination. At month 3, 6, 9 and 12 further treatments with intravitreal dexamethasone in combination with intravitreal ranibizumab are given if leakage is detected in fluorescein or indocyanine green (FLA or ICG) angiography, in case of further vision decrease or persistence of sub-/intraretinal fluid in OCT.
  Arms: Intravitreal dexamethasone and intravitreal ranibizumab
Drug: Intravitreal ranibizumab — Patients will receive intravitreal ranibizumab monotherapy (cohort 3). Study medications are initially given at the baseline visit. At each subsequent monthly follow-up visit, ranibizumab is administered if further visual deterioration or persistence of sub-/intraretinal fluid is detected in the examination
  Arms: Intravitreal ranibizumab

SUMMARY:
Age-related macular degeneration (AMD) is by far the most common disorder in the group of irreversible causes of visual disability. AMD leads to dysfunction and loss of photoreceptors in the central retina. Neovascular AMD (nAMD) affects visual function early in the disease process and severely compromises the highly developed functions of the macula, such as perception of details, central fixation, color vision, and reading ability. AMD-related visual impairment is associated with a loss of autonomy and quality of life. Current therapeutic approaches target vascular endothelial growth factor (VEGF), which has been identified as a main cytokine in the pathogenesis of nAMD. Ranibizumab, the fab-fragment of an antibody targeting VEGF is approved for the treatment of nAMD applied intravitreally in monthly intervals until the disease activity is stopped. However, a significant proportion of patients with nAMD suffer from persistent or recurring disease with the need of continuous anti-VEGF therapy over months and years, often leading to irreversible changes in the photoreceptor layer and the pigment epithelium.

Recent studies regarding the treatment of nAMD utilized different forms of therapies, combining photodynamic therapy with verteporfin (PDT) and ranibizumab, as well as therapeutic regimen containing steroids. Even though these studies did not provide evidence that combination therapies are superior to ranibizumab monotherapy, studies were only conducted with patients with previously untreated nAMD. Therefore, currently there is no alternative therapeutic approach for patients with recurrent or persistent form of nAMD after multiple treatments with ranibizumab monotherapy.

The purpose of this study is to assess the treatment effect of reduced fluence PDT and intravitreal ranibizumab versus intravitreal dexamethasone and ranibizumab versus intravitreal ranibizumab monotherapy in patients with persistent or recurrent choroidal neovascularization (CNV) due to AMD.

The investigators hypothesis is that these findings will offer new insights in the management of persistent or recurrent CNV secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years of age or older.
* Patients with persistent or recurrence subfoveal CNV lesion secondary to AMD
* Patients who have a BCVA score better than 20/400 in the study eye using ETDRS.
* At least 6 initial intravitreal ranibizumab monotherapy
* The initial intravitreal ranibizumab treatment performed within the last 6 - 12 months.

Exclusion Criteria:

* Any prior initial intravitreal treatment other than intravitreal ranibizumab.
* History of glaucoma filtration surgery, corneal transplant surgery or extracapsular extraction of cataract with phacoemulsification within six months preceding Visit 1, or a history of post-operative complications within the last 12 months preceding Visit 1 in the study eye (uveitis, cyclitis etc.).
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma mediation).
* Aphakia or absence of the posterior capsule in the study eye.
* Presence of a retinal pigment epithelial tear involving the macula in the study eye.
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either require medical or surgical intervention during the three-month study period to prevent or treat visual loss that might result from that condition.
* Active intraocular inflammation (grade trace or above) in the study eye.
* Any active infection involving eyeball adnexa.
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Other ocular conditions that require chronic concomitant therapy with systemic or topical ocular corticosteroids. Chronic concomitant therapy is defined as multiple doses taken daily for three or more consecutive days at any time within six months prior to screening or during the course of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
• Central visual function. | 12 months
• Changes of intraretinal morphologies (central retinal thickness). | 12 months

SECONDARY OUTCOMES:
• Measurement of levels of proteins in the ocular fluid. | 12 months
• Perfusion of the neovascular net (FLA and ICG). | 12 months
• Chorioretinal perfusion (ICG). | 12 months
• Retinal sensitivity (mfERG, Nidek MP-1 microperimetry) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, MD, Principal Investigator — Department of Ophthalmology, Medical University of Vienna
Locations (1):
- Department of Ophthalmology, Medical University of Vienna, Vienna, Austria